CLINICAL TRIAL: NCT06852313
Title: Save the Ovaries - Surgical Management of Simple Ovarian Cysts in Children and Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: Principal Investigator, Uchenna Kennedy, Principal Investigator, University Children's Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAVEOVPRO2025
Record Dates: First submitted 2025-02-19; First posted 2025-02-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cyst Benign
Keywords: Ovarian cyst; Laparoscopy; Child
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ovarian Cyst Deroofing (Experimental): The Ovarian cyst is deroofed with a specific, predefined technique: removal of a square of the cyst wall and overlying ovarian capsule of 16x16mm and suctioning of cyst contents.
  Interventions: Procedure: Laparoscopic ovarian cyst surgery
- Ovarian Cyst Enucleation (Experimental): The ovarian cyst is enucleated by complete removal of the cyst lining with preservation of surrounding ovarian tissue.
  Interventions: Procedure: Laparoscopic ovarian cyst surgery

INTERVENTIONS:
Procedure: Laparoscopic ovarian cyst surgery — Laparoscopic ovarian cyst surgery is any surgery with the goal of removal or drainage of an ovarian cyst. The exact surgical technique will be predefined by randomization.

SUMMARY:
The purpose of this study is to evaluate which operative technique should be used for managing simple ovarian cysts in girls and adolescents. The two techniques that are being compared are laparoscopic cyst enucleation and laparoscopic cyst deroofing. The investigators will assess the effect of both techniques on the ovarian reserve and the risk of cyst recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic simple cysts ≥ 4 cm with indication for surgical intervention
* Asymptomatic cysts ≥ 4 cm, with surgical indication due to persistence or increase in size
* Asymptomatic cysts ≥ 4 cm with other pathology as surgical indication, if known preoperatively
* Age 12 months - 18 years
* Parents/legal custodian and patient give consent, for patients unable to consent due to their health condition or developmental status they show no signs of unwillingness to participate
* Symptomatic simple cysts ≥ 4 cm with indication for surgical intervention on both ovaries (each ovary will count as one)

Exclusion Criteria:

* Neonatal ovarian cysts (age <12 months)
* Age >18 years
* Complex cysts (with solid components, e.g., Teratoma, risk or suspicion of malignancy)
* Paratubar/paraovarian cysts
* Medical reason that precludes cyst enucleation (e.g. severe coagulopathy)
* Neither signed informed consent form or inadequate german, french or english language skills to give informed consent

Ages: 1 Year to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-14 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative change of AMH level | 8 weeks
  Change in AMH level postoperatively compared to preoperative AMH levels (measured in pmol/L).

SECONDARY OUTCOMES:
Postoperative recurrence rate | 14 weeks
  Postoperative recurrence is defined as an ipsilateral asymptomatic cyst ≥ 4cm or a cyst of any size that requires a medical or surgical intervention due to symptoms at follow-up 6-8 weeks postoperatively.
  If the asymptomatic cyst is < 4cm, a second follow-up will be performed at 10-14 weeks postoperatively. Recurrence is then defined as ipsilateral asymptomatic cyst ≥ 4cm or a cyst of any size that requires a medical or surgical intervention due to symptoms.
  The outcome will be measured as "recurrence/no recurrence"

OTHER OUTCOMES:
Intraoperative complications | 2 weeks
  The investigators will describe any intraoperative complications.
Operative times | 2 weeks
  The investigators will measure the operative times in minutes for both techniques.
Postoperative ipsilateral ovarian volume on ultrasound | 14 weeks
  The postoperative ipsilateral ovarian volume will be calculated by ultrasound (Ovarian Volume: V (in ml) = long axis in cm x transversal axis x ap diameter x 0.5) and compared to published standard ovarian volumes in ml according to age.
Postoperative adnexal ratio | 14 weeks
  The adnexal ratio will be calculated by division of the volume of the affected ovary (in ml) with the volume of the unaffected ovary (in ml). If the adnexal ratio is <1 postoperatively, this can be a sign of postoperative volume loss.
Postoperative histology | 8 weeks
  The investigators will assess the histology of the cyst wall according to the following entities: functional cyst/ serous cystadenoma/ mucinous cystadenoma/ other entity.
Postoperative microscopic follicle count | 14 weeks
  The investigators will count the number of follicles that were removed on a representative sample of the surgical specimen, which will contain cyst wall +/- ovarian cortex.
Postoperative complications | 14 weeks
  Postoperative complications will be described by the Clavien-Madadi Classification.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Children's Hospital Basel, Basel
  - University Children's Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No